CLINICAL TRIAL: NCT00747734
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacology of MNRP1685A, a Human IgG1 Antibody, Administered Intravenously in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of MNRP1685A in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Disclosures Group, Genentech, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANP4509g
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Solid Cancers
Keywords: Neuropilin-1; NRP1; anti-NRP1; anti-angiogenic
MeSH Terms: interventions — vesencumab

INTERVENTIONS:
Drug: MNRP1685A — Escalating intravenous dose

SUMMARY:
This is a Phase I, first-in-human, open-label, dose-escalation study of MNRP1685A administered by IV infusion every 3 weeks in patients with locally advanced or metastatic solid tumors for whom standard therapy either does not exist or has proven to be ineffective or intolerable. This study will be conducted at up to three study centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Incurable, locally advanced, or metastatic solid malignancy that has progressed on, or failed to respond to, at least one prior regimen
* Evaluable or measurable disease per RECIST (in certain circumstances, prostate or ovarian cancer patients with non-measurable disease)

Exclusion Criteria:

* Inadequate hematologic or organ function
* Anti-cancer therapy within 4 weeks prior to initiation of study treatment
* Recent history of or current clinically significant gastrointestinal, cardiovascular or pulmonary disorders
* Any condition requiring full-dose anticoagulants, such as warfarin, heparin, or thrombolytics, or a filter of the inferior vena cava
* Active infection or autoimmune disease
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Length of study

SECONDARY OUTCOMES:
Total exposure (AUC) | Length of study
Maximum and minimum serum concentrations | Length of study
Clearance | Length of study
Volume of distribution | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Brachmann, M.D., Study Director — Genentech, Inc.